CLINICAL TRIAL: NCT01678820
Title: A Phase III, Randomized, Double-blind, Clinical Trial to Study the Efficacy and Safety of MK-0431D (a Fixed-dose Combination [FDC] of Sitagliptin and Simvastatin) for the Treatment of Patients With Type 2 Diabetes Mellitus (T2DM) With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: A Study of the Efficacy and Safety of MK-0431D (a Fixed-dose Combination of Sitagliptin and Simvastatin) for the Treatment of Participants With Type 2 Diabetes Mellitus (T2DM) With Inadequate Glycemic Control on Metformin Monotherapy (MK-0431D-266)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Merck terminated the study for business reasons in November 2013.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431D-266
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Simvastatin; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitagliptin/Simvastatin FDC (Experimental): Sitagliptin 100 mg/simvastatin 40 mg FDC plus placebo to sitagliptin plus placebo to simvastatin administered orally once daily in the evening for 16 weeks. Participants will continue on their stable pre-screening metformin dose and dosing regimen of >=1500 mg daily for the duration of the study. Participants may receive glimepiride 1 mg once daily or 2 mg once daily (may be up-titrated to 6 mg once daily) as rescue therapy.
  Interventions: Drug: Sitagliptin/Simvastatin FDC; Drug: Placebo to sitagliptin; Drug: Placebo to simvastatin; Drug: Metformin; Drug: Glimepiride
- Sitagliptin (Active Comparator): Sitagliptin 100 mg plus placebo to simvastatin plus placebo to sitagliptin/simvastatin FDC administered orally once daily in the evening for 16 weeks. Participants will continue on their stable pre-screening metformin dose and dosing regimen of >=1500 mg daily for the duration of the study. Participants may receive glimepiride 1 mg once daily or 2 mg once daily (may be up-titrated to 6 mg once daily) as rescue therapy.
  Interventions: Drug: Sitagliptin; Drug: Placebo to simvastatin; Drug: Placebo to Sitagliptin/Simvastatin FDC; Drug: Metformin; Drug: Glimepiride
- Simvastatin (Active Comparator): Simvastatin 40 mg plus placebo to sitagliptin plus placebo to sitagliptin/simvastatin FDC administered orally once daily in the evening for 16 weeks. Participants will continue on their stable pre-screening metformin dose and dosing regimen of >=1500 mg daily for the duration of the study. Participants may receive glimepiride 1 mg once daily or 2 mg once daily (may be up-titrated to 6 mg once daily) as rescue therapy.
  Interventions: Drug: Simvastatin; Drug: Placebo to sitagliptin; Drug: Placebo to Sitagliptin/Simvastatin FDC; Drug: Metformin; Drug: Glimepiride

INTERVENTIONS:
Drug: Sitagliptin/Simvastatin FDC — Sitagliptin 100 mg/Simvastatin 40 mg fixed-dose combination tablet
  Other Names: MK-0431D; Juvisync™; Juvicor®
  Arms: Sitagliptin/Simvastatin FDC
Drug: Sitagliptin — Sitagliptin 100 mg tablet
  Other Names: MK-0431; Januvia®; Tesavel®; Xelevia®; Ristaben®
  Arms: Sitagliptin
Drug: Simvastatin — Simvastatin 40 mg tablet
  Other Names: MK-0733; Zocor®
  Arms: Simvastatin
Drug: Placebo to sitagliptin — Matching placebo to sitagliptin 100 mg tablet
  Arms: Simvastatin; Sitagliptin/Simvastatin FDC
Drug: Placebo to simvastatin — Matching placebo to simvastatin 40 mg tablet
  Arms: Sitagliptin; Sitagliptin/Simvastatin FDC
Drug: Placebo to Sitagliptin/Simvastatin FDC — Matching placebo to sitagliptin 100 mg/simvastatin 40 mg FDC tablet
  Arms: Simvastatin; Sitagliptin
Drug: Metformin — Participants will continue on their stable, pre-screening metformin daily dose of >= 1500 mg for at least 12 weeks prior to randomization and during the study
  Other Names: Fortamet®; Glucophage®; Glucophage® XR; Glumetza®; Riomet®; Metgluco®; Glycoran®
Drug: Glimepiride — Following randomization, participants requiring glycemic rescue may receive open-label glimepiride initiated at a dose of 1 mg/day or 2 mg/day which may be up-titrated to 6 mg/day taken once daily with breakfast or the first main meal of the day.
  Other Names: Amaryl®; Glimy

SUMMARY:
The purpose of this study is to assess the efficacy and safety of sitagliptin/simvastatin fixed-dose combination (FDC) in participants with T2DM who have inadequate glycemic control while on metformin monotherapy. The primary hypothesis of this study is that after 16 weeks of therapy, the mean change from baseline in hemoglobin A1C (A1C) in participants treated with sitagliptin/simvastatin FDC is non-inferior compared to sitagliptin alone.

ELIGIBILITY:
Inclusion Criteria:

* has T2DM
* (1) Male; (2) female not of reproductive potential; or (3) female of reproductive potential who agrees to remain abstinent or use alone or in conjunction with their partner 2 methods of contraception to prevent pregnancy during the study and for 14 days after the last dose of study drug
* is currently on metformin monotherapy at a daily dose of at least 1500 mg for at least 10 weeks
* is not on a lipid-lowering agent for at least 6 weeks prior to entering the study

Exclusion Criteria:

* has history of type 1 diabetes mellitus (T1DM), or a history of ketoacidosis or possibly has T1DM
* has been on a thiazolidinedione (TZD) within the previous 16 weeks
* has been treated with a statin or other lipid-lowering agent (including over-the-counter [OTC] supplements) within the previous 6 weeks
* currently participating in or has participated in another clinical study within the past 12 weeks
* intends to consume >1.2 liters of grapefruit juice daily during the study
* is on or likely to require treatment for at least 2 consecutive weeks or repeated courses of corticosteroids (inhaled, nasal and topical corticosteroids are permitted)
* intolerance or hypersensitivity to sitagliptin, simvastatin, metformin or glimepiride
* is on a weight loss program and not in the maintenance phase or has started a weight loss medication or has undergone bariatric surgery in the previous 12 months
* has undergone a surgical procedure in the past 4 weeks or planned major surgery during the study
* has symptomatic hyperglycemia that requires immediate initiation, adjustment, or addition of antihyperglycemic therapy
* has a history of myopathy or rhabdomyolysis with any statin
* has cardiovascular disease, a diagnosis of congestive heart failure, or uncontrolled high blood pressure
* has a history of active liver disease
* has chronic progressive neuromuscular disorder, human immunodeficiency virus (HIV), hematological disorder, or uncontrolled endocrine or metabolic disease
* is currently being treated for hyperthyroidism or is on thyroid hormone therapy and has not been on a stable dose for at least 6 weeks
* has a history of malignancy in the previous 5 years (excluding adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer)
* is pregnant or breast feeding, or is expecting to conceive or donate eggs during the course of the study, including 14 days after the last dose of study drug
* is a user of recreational or illicit drugs or has had a recent history of drug abuse
* consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2013-11-01 (Actual); Study Completion 2013-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431D-266&kw=0431D-266&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants randomized population.
Groups:
- Sitagliptin/Simvastatin FDC: Sitagliptin 100 mg/simvastatin 40 mg FDC plus placebo to sitagliptin plus placebo to simvastatin administered orally once daily in the evening. Participants will continue on their stable pre-screening metformin dose and dosing regimen of >=1500 mg daily for the duration of the study. Participants may receive glimepiride 1 mg once daily or 2 mg once daily (may be up-titrated to 6 mg once daily) as rescue therapy.
- Sitagliptin: Sitagliptin 100 mg plus placebo to simvastatin plus placebo to sitagliptin/simvastatin FDC administered orally once daily in the evening. Participants will continue on their stable pre-screening metformin dose and dosing regimen of >=1500 mg daily for the duration of the study. Participants may receive glimepiride 1 mg once daily or 2 mg once daily (may be up-titrated to 6 mg once daily) as rescue therapy.
- Simvastatin: Simvastatin 40 mg plus placebo to sitagliptin plus placebo to sitagliptin/simvastatin FDC administered orally once daily in the evening. Participants will continue on their stable pre-screening metformin dose and dosing regimen of >=1500 mg daily for the duration of the study. Participants may receive glimepiride 1 mg once daily or 2 mg once daily (may be up-titrated to 6 mg once daily) as rescue therapy.
Period: Overall Study
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Started | 100 | 99 | 100
Treated With Double-blind Study Drug | 100 | 97 | 98
Completed | 38 | 36 | 43
Not Completed | 62 | 63 | 57
Not completed — Study Terminated by Sponsor | 45 | 43 | 43
Not completed — Withdrawal by Subject | 2 | 5 | 2
Not completed — Protocol Specified Criteria | 2 | 3 | 1
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Lost to Follow-up | 7 | 2 | 2
Not completed — Non-compliance with study drug | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Violation | 4 | 5 | 4
Not completed — Not treated with double-blind study drug | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants randomized population. Study specific baseline characteristics include all randomized participants with data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin | Total
Number analyzed (Participants) | 100 | 99 | 100 | 299
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (10.2) | 54.2 (10.3) | 54.9 (10.0) | 54.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 52 | 49 | 146
  Male | 55 | 47 | 51 | 153
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] | 8.16 (0.94) | 8.15 (1.09) | 8.22 (1.19) | 8.18 (1.08)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 169.9 (42.3) | 175.9 (48.6) | 175.7 (49.3) | 173.8 (46.8)
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 106.5 (26.7) | 103.9 (24.2) | 100.9 (22.0) | 103.7 (24.4)
Total cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 189.3 (30.9) | 187.7 (29.6) | 183.5 (28.4) | 186.8 (29.6)
Apolipoprotein B (Apo B) [Mean (Standard Deviation); unit: mg/dL] — Sitagliptin, n=95; Total, n=295
  mg/dL | 97.8 (19.0) | 95.4 (19.0) | 94.1 (17.2) | 95.8 (18.4)
Non high-density lipoprotein cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Sitagliptin, n=97; Total, n=297
  mg/dL | 141.7 (30.9) | 139.5 (29.9) | 136.5 (27.1) | 139.2 (29.3)
Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] | 177.4 (101.2) | 180.8 (119.1) | 184.2 (118.6) | 180.8 (112.9)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 47.6 (11.3) | 48.2 (12.1) | 47.0 (11.2) | 47.6 (11.5)
Very low-density lipoprotein cholesterol (VLDL-C) [Mean (Standard Deviation); unit: mg/dL] — Sitagliptin, n=97; Total, n=297
  mg/dL | 35.4 (18.8) | 35.8 (20.4) | 35.7 (18.8) | 35.6 (19.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 16 (Sitagliptin/Simvastatin FDC vs. Sitagliptin)
Description: A1C is measured as percent. Thus, this change from baseline reflects the Week 16 A1C percent minus the Week 0 A1C percent. This primary outcome measure only includes results for sitagliptin/simvastatin FDC vs. sitagliptin. Results for simvastatin are presented below under secondary outcome measures.
Time Frame: Baseline and Week 16
Population: Full analysis set (FAS) population defined as all randomized participants who took at least one dose of study drug and had at least one measurement for the analysis of this outcome measure (baseline or subsequent to the first dose of study drug).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin
Number analyzed (Participants) | 100 | 97
Percent | -0.41 [-0.64 to -0.17] | -0.59 [-0.83 to -0.36]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; p = 0.267, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = 0.19, 95% CI 2-sided [-0.14 to 0.52]

2. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: Excludes data after rescue therapy. Adverse event is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product.
Time Frame: Up to 16 weeks for non-serious AEs, up to 18 weeks for serious AEs
Population: All participants as treated population defined as all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 97 | 98
Participants | 13 | 13 | 17
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; Difference in percents = -0.4, 95% CI 2-sided [-10.2 to 9.3] — Based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; Difference in percents = -4.3, 95% CI 2-sided [-14.7 to 5.8] — Based on Miettinen & Nurminen method

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 2
Time Frame: Up to 16 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 97 | 98
Participants | 2 | 1 | 2

4. Secondary Outcome: Change From Baseline in A1C at Week 16 (Sitagliptin/Simvastatin FDC vs. Simvastatin)
Description: A1C is measured as percent. Thus, this change from baseline reflects the Week 16 A1C percent minus the Week 0 A1C percent. This primary outcome measure only includes results for sitagliptin/simvastatin FDC vs. simvastatin. Results for sitagliptin are presented above under primary outcome measures.
Time Frame: Baseline and Week 16
Population: FAS population defined as all randomized participants who took at least one dose of study drug and had at least one measurement for the analysis of this outcome measure (baseline or subsequent to the first dose of study drug).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin/Simvastatin FDC | Simvastatin
Number analyzed (Participants) | 100 | 98
Percent | -0.41 [-0.64 to -0.17] | 0.21 [-0.02 to 0.45]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = -0.62, 95% CI 2-sided [-0.95 to -0.28]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 16
Description: Change from baseline reflects the Week 16 value minus the Week 0 value.
Time Frame: Baseline and Week 16
Population: FAS population defined as all randomized participants who took at least one dose of study drug and who had at least one measurement for the analysis of this outcome measure (baseline or subsequent to the first dose of study drug).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 97 | 98
mg/dL | -7.9 [-21.0 to 5.2] | -9.6 [-23.4 to 4.1] | 21.3 [7.9 to 34.7]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; p = 0.856, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = 1.7, 95% CI 2-sided [-17.1 to 20.6]
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; p = 0.002, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = -29.2, 95% CI 2-sided [-47.9 to -10.6]

6. Secondary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Week 16
Description: Percent change from baseline was calculated as the Week 16 value minus the Week 0 value, divided by the Week 0 value ×100%.
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 97 | 98
Percent change | -21.6 [-32.3 to -10.8] | 4.0 [-6.9 to 14.9] | -26.9 [-37.5 to -16.3]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = -25.6, 95% CI 2-sided [-35.6 to -15.6]
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; p = 0.286, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = 5.3, 95% CI 2-sided [-4.5 to 15.2]

7. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 97 | 98
Percent change | -18.4 [-26.6 to -10.2] | -0.4 [-8.6 to 7.9] | -18.4 [-26.4 to -10.4]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = -18.1, 95% CI 2-sided [-24.2 to -12.0]
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; p = 0.990, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = -0.0, 95% CI 2-sided [-6.0 to 6.0]

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 94 | 98
Percent change | -16.9 [-27.0 to -6.8] | 3.3 [-7.1 to 13.7] | -19.8 [-30.0 to -9.6]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = -20.2, 95% CI 2-sided [-28.3 to -12.2]
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; p = 0.469, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = 2.9, 95% CI 2-sided [-5.0 to 10.7]

9. Secondary Outcome: Percent Change From Baseline in Non-high Density Lipoprotein Cholesterol (Non-HDL-C) at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 96 | 98
Percent change | -23.9 [-33.9 to -13.9] | 0.6 [-9.5 to 10.7] | -24.2 [-34.0 to -14.4]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; p < 0.001, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = -24.4, 95% CI 2-sided [-32.6 to -16.3]
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; p = 0.937, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = 0.3, 95% CI 2-sided [-7.7 to 8.3]

10. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 97 | 98
Percent change | -20.4 [-51.9 to 11.1] | -4.9 [-39.5 to 29.7] | -10.1 [-52.1 to 31.9]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; p = 0.068, Robust regression; Using M-estimation with treatment, region, and a covariate for baseline triglycerides (mg/dL). Missing data were imputed by multiple imputations; Difference in estimated means = -15.5, 95% CI 2-sided [-32.2 to 1.2]
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; p = 0.365, Robust regression; [statistical method as in outcome 10, analysis 1]; Difference in estimated means = -10.3, 95% CI 2-sided [-33.6 to 13.0]

11. Secondary Outcome: Percent Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 97 | 98
Percent change | 2.5 [-2.7 to 7.8] | 2.0 [-3.3 to 7.4] | 2.1 [-3.0 to 7.3]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; p = 0.857, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = 0.5, 95% CI 2-sided [-4.8 to 5.8]
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; p = 0.879, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = 0.4, 95% CI 2-sided [-4.8 to 5.6]

12. Secondary Outcome: Percent Change From Baseline in Very Low-density Lipoprotein Cholesterol (VLDL-C) at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 96 | 98
Percent change | -17.5 [-33.8 to -1.2] | 12.9 [-4.2 to 29.9] | -2.2 [-18.9 to 14.5]
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; p = 0.004, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = -30.4, 95% CI 2-sided [-51.0 to -9.7]
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; p = 0.141, Longitudinal Data Analysis Model; Based on a longitudinal model including terms for region, treatment, time, and the interaction of time by treatment; Difference in least squares means = -15.3, 95% CI 2-sided [-35.8 to 5.1]

13. Secondary Outcome: Percentage of Participants With A1C Level <7% at Week 16
Description: Percentage of participants achieving glycemic goal (A1C <7%) after 16 weeks of treatment. Data as observed.
Time Frame: Week 16
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Number analyzed (Participants) | 100 | 97 | 98
Percentage of participants | 29.9 | 29.6 | 17.6
Statistical Analysis 1: Comparison: Sitagliptin/Simvastatin FDC vs Sitagliptin; Test type: Superiority or Other; Difference in percents = 0.3, 95% CI 2-sided [-12.2 to 12.9] — Based on Miettinen & Nurminen method. Missing data were imputed by multiple impuattions
Statistical Analysis 2: Comparison: Sitagliptin/Simvastatin FDC vs Simvastatin; Test type: Superiority or Other; Difference in percents = 12.3, 95% CI 2-sided [0.7 to 24.0] — Based on Miettinen & Nurminen method. Missing data were imputed by multiple imputations

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Description: All participants as treated population defined as all randomized participants who received at least one dose of study drug. Serious adverse events include data after rescue therapy and non-serious adverse events exclude data after rescue therapy.
Arm/Group | Sitagliptin/Simvastatin FDC | Sitagliptin | Simvastatin
Serious Adverse Events (participants affected / at risk) | 1/100 | 0/97 | 1/98
Other Adverse Events (participants affected / at risk) | 0/100 | 0/97 | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Simvastatin FDC (N=100) | Sitagliptin (N=97) | Simvastatin (N=98)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated for business reasons in November 2013.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.